CLINICAL TRIAL: NCT03868423
Title: Phase II Study of Brigatinib for Advanced Solid Cancers Harboring Genomic Alterations in ALK (Excluding Lung) and ROS1 Oncogenes
Brief Title: Brigatinib in Treating Patients With ALK and ROS1 Gene Alterations and Locally Advanced or Metastatic Solid Cancers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI decision
Sponsor: Sameek Roychowdhury (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Sameek Roychowdhury, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-17060; NCI-2017-01394 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016058 (NIH)
Record Dates: First submitted 2019-02-04; First posted 2019-03-11 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Advanced Malignant Neoplasm; ALK Fusion Protein Expression; ALK Gene Amplification; ALK Gene Mutation; Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Neoplasm in the Central Nervous System; Metastatic Malignant Solid Neoplasm; ROS1 Fusion Positive; ROS1 Gene Amplification; ROS1 Gene Mutation
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — brigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (brigatinib) (Experimental): Patients receive brigatinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brigatinib; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Brigatinib — 90 mg orally QD for 7 days followed by 180 mg orally QD continuously thereafter. One cycle of therapy will consist of 28 days of treatment.
  Other Names: Alunbrig; AP 26113; AP-26113; AP26113
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well brigatinib works in treating patients with ALK and ROS1 gene alterations and solid cancers that have spread to nearby tissue and lymph nodes or other places in the body. Brigatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the overall response rate (ORR) of brigatinib in patients with advanced solid tumors harboring genomic alterations in ALK (excluding lung) and ROS1 (all solid tumors).

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of brigatinib in patients with advanced solid tumors harboring genomic alterations in ALK (excluding lung) and ROS1 (all solid tumors).

II. To assess progression free survival (PFS) and overall survival (OS) in patients with advanced ALK or ROS1 mutated solid tumors treated with brigatinib.

III. To assess sensitivity and durability of response to brigatinib in different solid tumor types.

IV. To assess the role of intertumoral and intratumoral heterogeneity in the development of resistance to brigatinib.

V. To identify candidate genomic (including circulating tumor deoxyribonucleic acid [DNA]) and proteomic biomarkers of tumor sensitivity and resistance to brigatinib using high-throughput approaches (exome, transcriptome, reverse phase protein array [RPPA]).

TERTIARY OBJECTIVES:

I. Correlation of brigatinib exposure with efficacy and safety. II. Correlation of tumor and plasma biomarkers with brigatinib efficacy and safety.

OUTLINE:

Patients receive brigatinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumors
* Patients must have activating genomic alterations in ALK or ROS1 (mutations, fusions or amplifications) by any validated Clinical Laboratory Improvement Act (CLIA)-certified molecular testing (fluorescence in situ hybridization [FISH], polymerase chain reaction [PCR] or next-generation sequencing [NGS] data are acceptable); CLIA validated results from other institutions and commercial diagnostic labs (e.g. Foundation Medicine) are also acceptable
* Patients with progressive disease on any previous therapy including crizotinib and other ALK tyrosine kinase inhibitors (TKIs), chemotherapy or immunotherapy
* Patients with locally advanced or metastatic solid tumors who have received no previous therapy of any kind (i.e. first-line therapy) are eligible
* Patients with brain metastases or metastases elsewhere within the central nervous system (CNS) are eligible for study; patients must be neurologically stable and asymptomatic
* Patients with tumor suitable for biopsy (as assessed by trained specialists in interventional radiology) and medically fit to undergo a biopsy or surgical procedure will have mandatory pre-treatment tumor biopsy or sampling; however, if patients do not have a tumor suitable for biopsy but have another tissue (preferably progressive metastatic site) available for molecular evaluation this will be acceptable
* Patients with solid tumors must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1; Note: previously irradiated lesions may not be used for target lesions; unless there is unambiguous radiological progression after radiotherapy; brain lesions may not be used as target lesions if they were: 1) previously treated with whole brain radiation therapy (WBRT) within 3 months, or 2) previously treated by stereotactic radiosurgery (SRS) or surgical resection
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy of greater than 3 months
* Patients with multiple malignancies remain eligible
* Patients with an inherited cancer syndrome or a medical/family history suggestive of an inherited cancer syndrome remain eligible
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and through 4 months after the end of treatment; for women of childbearing potential, a negative pregnancy test must be documented prior to registration
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 10 g/dL
* Platelet count >= 75,000/mcL
* Total bilirubin =< 1.5 x upper limit of normal (ULN), unless due to Gilbert?s syndrome (< 5 if metastatic involvement of the liver)
* Serum lipase =< 1.5 x ULN
* Serum amylase =< 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Left ventricular ejection fraction (LVEF) >= 50% by echocardiogram or multi-gated acquisition (MUGA)
* Normal QT interval on screening electrocardiogram (ECG), defined as QT interval corrected of =< 450 ms in males or =< 470 ms in females
* Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockroft-Gault formula) >= 60 mL/min OR 24-hour urine creatinine clearance >= 60 mL/min
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with hematological malignancies
* Patients with ALK positive (+) lung cancer
* Major surgery (e.g. thoracic, abdominal, vascular, neurosurgery) within 30 days prior to registration on study
* Pregnant women or mothers who are breastfeeding
* Patients who are incarcerated
* Patients who have a history or the presence at baseline of pulmonary interstitial disease or drug-related pneumonitis, or radiation pneumonitis
* Patients who have a known history of human immunodeficiency virus (HIV); testing not required in the absence of history
* Patients with history of clinically significant bleeding disorder or history of active significant gastrointestinal (GI) bleeding within 3 months of first dose of brigatinib
* Patients who have malabsorption syndrome or other GI illness or condition that could affect oral absorption of the study drug
* History of allergic or suspected hypersensitivity reactions attributed to compounds of similar chemical or biologic composition to brigatinib
* Patients with history of clinically significant atrial arrhythmias (requiring any anti-arrhythmic therapy or as determined by the treating physician) or any history of ventricular arrhythmias
* Patients who have significant, uncontrolled or active cardiovascular disease, including but not restricted to the following:

  * Myocardial infarction (MI) within 6 months prior to first dose of brigatinib
  * Unstable angina (UA) within 6 months prior to first use
  * Decompensated congestive heart failure within 6 months prior to first dose
  * Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months prior to first dose
* Clinically significant, uncontrolled intercurrent illness including, but not limited to:

  * Symptomatic or active infection requiring intravenous (IV) antibiotics
  * Psychiatric illness and/or social situations that would limit compliance with completion of study requirements
* Patients on medications known to be associated with torsades de pointes
* Patients who have uncontrolled hypertension; patients with hypertension should be under treatment on study entry to control blood pressure
* Patients who have received cytotoxic chemotherapy, investigational agents, or radiation within 14 days, except stereotactic radiosurgery (SRS) or stereotactic body radiosurgery
* Patients who have received monoclonal antibodies or had major surgery within 30 days of the first dose of brigatinib
* Patients who have not recovered (=< Common Terminology Criteria for Adverse Events [CTCAE] grade 1) from adverse events (with the exception of alopecia) due to agents administered more than 4 weeks earlier
* Patients with symptomatic CNS metastases that are neurologically unstable or require increasing dose of corticosteroids
* Patients with current spinal cord compression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate assessed per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 52 weeks
  Response for tumors will be assessed using the RECIST 1.1 criteria (using computed tomography scans or calipers by clinical exam) where response will be defined as a partial or complete response. Will be calculated with 95% binomial confidence intervals for the estimate of the proportion of responses.

SECONDARY OUTCOMES:
Confirmed objective response rate (ORR) | Up to 52 weeks
  Will be assessed by central independent review committee per RECIST version 1.1.
Time to response | Up to 52 weeks
  Will be evaluated.
Duration of response | From the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 52 weeks
  Will be evaluated.
Time on treatment | Up to 52 weeks
  Will be evaluated.
Disease control rate | Up to 52 weeks
  Will be assessed by RECIST version 1.1.
Incidence of adverse events assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 52 weeks
  Frequency and severity of adverse events and tolerability of the regimen will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Overall survival | From treatment initiation to death due to any cause, assessed up to 52 weeks
  Kaplan-Meier curves will be used to estimate the survival distributions of overall survival.
Progression-free survival | From the date of study registration to the date of event (ie, death and/or disease progression) or the date of last follow-up if no event has occurred, up to 52 weeks
  Kaplan-Meier curves will be used to estimate the survival distributions of progression-free survival.
Clinical benefit rate | 6 months
  Will be calculated by the number of patients who have achieve a response and/or are progression-free and alive at 6 months divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for clinical benefit rate will be calculated.
Rate of participation of those screened and identified with the eligible genetic alterations | Up to 52 weeks
  The logistical aspects of the trial will be evaluated and summarized. Disease group-specific outcomes will also be summarized and described, although we will not be powered for any formal evaluation within a disease or histology subset.
Rate of enrollment of those screened and identified with the eligible genetic alterations | Up to 52 weeks
  The logistical aspects of the trial will be evaluated and summarized. Disease group-specific outcomes will also be summarized and described, although we will not be powered for any formal evaluation within a disease or histology subset. Genes will be evaluated in aggregate from whole exome and transcriptome sequencing.

OTHER OUTCOMES:
Brigatinib exposure | Up to 52 weeks
  Brigatinib exposure will be compared to RECIST measurements and adverse events measured using CTCAE v4.
Correlative gene and protein markers | Up to 52 weeks
  Correlative and protein markers will be summarized univariately in a quantitative manner and also summarized by clinical outcome group (e.g. response vs. no response). Graphical analyses will be largely used to assess potential patterns and relationships; e.g. side-by-side boxplots to assess differences in continuous marker levels between those with vs. without the clinical improvement (e.g. response versus no response). Will correlate with efficacy and safety.

CONTACTS AND LOCATIONS:
Overall Officials: Sameek Roychowdhury, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu